CLINICAL TRIAL: NCT00593372
Title: Treatment of Language and Memory in Patients With Alzheimer's Disease: A Comparison Between Drug Therapy and Drug Therapy Plus Behavioral Intervention
Brief Title: Treatment of Language and Memory in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: g1-10532-03-07
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2010-07-20 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Memory; Treatment
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Drug Plus Behavioral Therapy
  Interventions: Behavioral: Spaced Retrieval Training
- II (No Intervention): Drug Therapy Only

INTERVENTIONS:
Behavioral: Spaced Retrieval Training — Increasing time to remember important information.
  Arms: I

SUMMARY:
The purpose of this study is to collect data on the effects of behavioral interventions for memory and communication deficits in persons taking cholinesterase inhibitors compared with the effects of cholinesterase inhibitors alone. Initial testing will include a written case history, tests of communication skills, and interviews with the participants, family, and staff caregivers to help select potential goals for treatment. Participants will be randomly selected to participate in Group A (control) or Group B (intervention). Group A will use a Caregiver Checklist for eight weeks to identify any increase or decrease in the occurrence of the identified communication deficits. Group B will have 16 treatment sessions by a Speech Language Pathologist during the eight-week period. A post test will be administered to all participants.

DETAILED DESCRIPTION:
Patients with dementia suffer from a variety of cognitive-linguistic deficits, including attention, orientation, memory, anomia, and pragmatics. Behavioral treatment of these deficits falls within the domain of speech-language pathology. While no efficacy studies have emerged to demonstrate the benefit of speech-language therapy for individuals who suffer Alzheimer's disease (AD), data are emerging which support the positive effects of memory and communication intervention in this population. Phase I and Phase II investigations are beginning to provide evidence that such intervention should focus on the development of innovative strategies to help patients compensate for the disabilities resulting from the disease rather than on traditional rehabilitation of impairment. The benefits of cholinesterase inhibitors for improving cognitive function in persons with AD have been demonstrated, and data continue to emerge on specific drugs and specific changes in cognitive processes. The purpose of the proposed investigation would be to collect pilot data on the effects of behavioral intervention for memory and communication deficits in conjunction with cholinesterase inhibitors, as compared with the effects of cholinesterase inhibitors used in isolation. Participants will be individuals with AD who are recruited from the Alzheimer's Disease Center at The University of Arkasas for Medical Sciences Medical Center. All participants will be taking cholinesterase inhibitors, and half of all participants will be randomly selected to receive intervention by a speech-language pathologist. Intervention will consist of 16 treatment sessions (one hour each) over a two month period and will focus on strategies for enhancing memory and functional communication.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's Disease (middle stage)

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary H McCullough, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- UAMS Medical Center, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Spaced Retrieval Therapy: Participants continue on current medication but participate in spaced retrieval memory training, as well.
- Continuing Medication Only: Participants continue on current medication and are assessed at beginning and end of study duration.
Period: Overall Study
Arm/Group | Spaced Retrieval Therapy | Continuing Medication Only
Started | 8 (Eight enrolled in behavioral treatment.) | 3 (Three evaluated but only maintained medical treatment.)
Completed | 8 (Eight completed behavioral treatment.) | 3 (Three evaluated and completed protocol.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spaced Retrieval Therapy | Continuing Medication Only | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (5) | 72 (3) | 72 (6)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Memory Tasks Completed Over Study Period.
Description: Successful memory tasks are those memory tasks (such as "where do I keep my keys") that participants are able to consistently respond to.
Time Frame: 8 weeks
Measure: Number; unit: memory tasks
Arm/Group | Spaced Retrieval Therapy | Continuing Medication Only
Number analyzed (Participants) | 8 | 3
memory tasks | 5 | 0

2. Secondary Outcome: Change on Mini-Mental State Examination
Time Frame: End of Study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Spaced Retrieval Therapy | Continuing Medication Only
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3

LIMITATIONS AND CAVEATS:
Recruitment of participants was the major limitation of the trial. Alzheimer's patients at facility were asked to participate in so many studies, that participation in this one was challenging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes